CLINICAL TRIAL: NCT06405698
Title: A Randomized Comparison Between Perforator Flap vs Perforator Plus Flap in Myelomeningocele Defect Repair
Brief Title: Role of Perforator Flaps in Back Defects Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed elsayed tawfik, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: flaps in myelomeningiocele
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Myelomeningocele
Keywords: myelomeningocele; perforator flaps; infants
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- closure of the myelomeningocele defect by perforator flap. (Experimental): fifteen patient with myelomeningocele defect
  Interventions: Procedure: surgical closure of myelomeningocele defects by perforator flaps
- closure of the myelomeningocele defect by perforator plus flap . (Experimental): fifteen patient with myelomeningocele defect
  Interventions: Procedure: surgical closure of myelomeningocele defects by perforator-plus flaps

INTERVENTIONS:
Procedure: surgical closure of myelomeningocele defects by perforator flaps — closure of myelomeningocele defect by perforator island flap after complete incision of the flap all around based on perforator vessel .
  Arms: closure of the myelomeningocele defect by perforator flap.
Procedure: surgical closure of myelomeningocele defects by perforator-plus flaps — closure of myelomeningocele defect by perforator-plus island flap harvesting leaving skin bridge connecting to the flap and dissection of the perforator vessel
  Arms: closure of the myelomeningocele defect by perforator plus flap .

SUMMARY:
evaluation of perforator flaps versus perforator plus flaps

DETAILED DESCRIPTION:
One of the neural tube defects, myelomeningocele, is a congenital anomaly developing in the fourth gestational week. It is characterized by insertion of neural elements into a pouch floored by meninx through a vertebral defect.

The aetiology is multifactorial. causes are genetic properties, geographic factors, and deficiency of folic acid.

Meningomyelocele incidence range between 1 and 2/1000 live births. The defect location can reside anywhere between the cervical region and the sacrum.

surgical closure of the defect is performed to prevent cerebrospinal fluid leakage and central nervous system infections. it is a combined work between neurosurgery and plastic surgery. Fascial turnover flaps, muscle flaps, local fasciocutaneous flaps.

With the emerging concepts of perforator flaps in the last three decades, the reconstruction of myelomeningocele defects has completely changed since the anatomy of the dorsal intercostal artery perforators (DIAP) and lumbar artery perforators(LAP) has been fully studied.

Despite utilizing perforator flaps having greatly improved the outcome of myelomeningocele reconstruction, venous compromise remained a major concern associated with complications.

By preserving, the perforator vessels and minimizing the amount of tissue that is removed, the Perforator Plus technique can improve blood flow and decrease the risk of venous congestion.

Preoperative perforator mapping may be executed by a multitude of diagnostic modalities. Hand-held Doppler (HHD), color-coded duplex sonography (CCDS), computed tomography angiography (CTA), magnetic resonance angiography (MRA) and others may be applied.

Systematic reviews of the literature revealed that CCDS has the highest sensitivity and positive predictive value to identify perforators for flaps.

ELIGIBILITY:
Inclusion Criteria:

* infants up to one year,
* dorso-lumbar myelomeningocele.
* moderate to large myelomeningocele defects. (25 - 39 cm2 ) .

Exclusion Criteria:

* cervical myelomeningocele
* very large defects (more than 40 cm2 )
* preterm newborn patients.
* hematological disease
* any problem against prone position of the patient

Ages: 2 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
changing complication rate | baseline and 3 months
  evaluate of different flaps modalities in back defects closure
changing hospital stay time | baseline and one month

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud Abdelaal, doctor, Study Director — professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isik D, Tekes L, Eseoglu M, Isik Y, Bilici S, Atik B. Closure of large myelomeningocele defects using dorsal intercostal artery perforator flap. Ann Plast Surg. 2011 Aug;67(2):159-63. doi: 10.1097/SAP.0b013e3181f3e0cf. PMID 21301309
- [Background] Cologlu H, Ozkan B, Uysal AC, Cologlu O, Borman H. Bilateral propeller flap closure of large meningomyelocele defects. Ann Plast Surg. 2014 Jul;73(1):68-73. doi: 10.1097/SAP.0b013e31826caf5a. PMID 24918736
- [Background] Basterzi Y, Tenekeci G. Dorsal Intercostal Artery Perforator Propeller Flaps: A Reliable Option in Reconstruction of Large Meningomyelocele Defects. Ann Plast Surg. 2016 Apr;76(4):434-7. doi: 10.1097/SAP.0000000000000417. PMID 26010351
- [Background] Kehrer A, Heidekrueger PI, Lonic D, Taeger CD, Klein S, Lamby P, Sachanadani NS, Jung EM, Prantl L, Batista da Silva NP. High-Resolution Ultrasound-Guided Perforator Mapping and Characterization by the Microsurgeon in Lower Limb Reconstruction. J Reconstr Microsurg. 2021 Jan;37(1):75-82. doi: 10.1055/s-0040-1702162. Epub 2020 Feb 28. PMID 32110822